CLINICAL TRIAL: NCT06285123
Title: Implementing the COMFORT Guidelines for Postpartum Pain Management: A Statewide Quality Improvement Project in the Obstetrics Initiative
Brief Title: Implementing the COMFORT Guidelines for Postpartum Pain Management
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle H. Moniz, Principal Investigator, University of Michigan
Other Study IDs: HUM00248235 and HUM00248331; 1U01FD007803-01 (FDA)
Record Dates: First submitted 2024-02-01; First posted 2024-02-29 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Postpartum Pain; Opioid Stewardship; Maternity Care; Obstetric Care
Keywords: Quality Improvement; Clinical Practice Guidelines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Responders
  Interventions: Behavioral: REP
- Non-Responders REP
  Interventions: Behavioral: REP
- Non-Responders REP/Facilitation
  Interventions: Behavioral: REP; Behavioral: Facilitation

INTERVENTIONS:
Behavioral: REP — REP is a bundle of strategies designed to help hospitals implement an evidence-based clinical practice. REP's core components include 1) user-friendly "packaging" of the clinical guidance, 2) structured clinician training, 3) performance feedback, and 4) brief technical assistance.
Behavioral: Facilitation — Facilitation is a process of interactive problem-solving via a supportive consultation relationship. Facilitation is delivered by an expert who meets regularly with site quality improvement leaders to support interactive problem-solving to address local barriers and unanticipated implementation challenges. In contrast to the group-based, brief technical assistance in REP, facilitation is individualized consultation with the site clinical champion that generates highly customized, local solutions that can potentially be sustained by the local providers and champions.
  Groups: Non-Responders REP/Facilitation

SUMMARY:
A new national clinical practice guideline (CPG) for pain management after childbirth aims to mitigate peripartum opioid-related risks without compromising or exacerbating existing inequities in pain management in the United States. Standard dissemination approaches are often insufficient to change clinical practice-more active implementation efforts are generally required. Replicating Effective Programs (REP) is a theory-driven implementation intervention that is publicly available and highly scalable, but REP alone may be insufficient for effectively embedding the CPG across all maternity sites. For sites needing more support, REP can be augmented with facilitation (e.g., individualized consultation with site champions to overcome local barriers to CPG adoption, "Enhanced-REP" [E-REP]). Because E-REP is more expensive and difficult to scale than REP, it is essential to identify those settings where REP alone is effective versus those where REP may need augmentation, but this has not been evaluated in maternity contexts. Our objective is to determine the effect of a new postpartum pain management CPG, as implemented by REP and E-REP, on postpartum opioid prescribing (primary outcome: rate and amount of opioid prescribed within three days of childbirth), overall, by hospital, and among key subgroups.

This is a non-responder randomized trial within the Obstetrics Initiative (OBI), a perinatal collaborative quality initiative funded by Blue Cross Blue Shield of Michigan that includes 68 member hospitals serving more than 120,000 postpartum people over an approximately 15-month study time period. Hospitals not initially responding to REP (defined by performance below the top 15th percentile of all OBI hospitals for a) inpatient order for opioid-sparing postpartum pain management, [e.g., scheduled acetaminophen and ibuprofen], or b) amount of opioid prescribed at discharge, or c) provision of non-medication pain management interventions) will be allocated, via block randomization, to either continue REP vs. augment REP with facilitation (E-REP).

The primary analysis will evaluate the rate of postpartum opioid-sparing prescribing metrics at the time of discharge (primary outcome) and opioid prescription refills and high-risk prescribing (secondary outcomes) before and after CPG implementation with REP, using interrupted time series analyses. Inequities in outcomes by patient, procedure, prescriber, and hospital factors will be evaluated. Exploratory analyses will examine temporal trends in patient-reported outcomes. The effects of continued REP vs. E-REP among non-responder sites will also be examined. Finally, implementation outcomes will be characterized using clinician and patient surveys and qualitative methods.

DETAILED DESCRIPTION:
This record is for one observational study with two unique institutional identifiers (HUM00248235 and HUM00248331). Because outcome measure 6 met a different exemption criteria than the other outcome measures, the IRB issued two unique identifiers, although both identifiers are for the same study. To avoid creating duplicate records, and to accurately represent this as a single study, only one record was registered in the ClinicalTrials.gov system.

ELIGIBILITY:
Inclusion Criteria:

-All hospitals fully participating in the Obstetrics Initiative (OBI), a Blue Cross Blue Shield of Michigan (BCBSM)-funded collaborative of Michigan hospitals dedicated to maternity care quality improvement.

Exclusion Criteria:

-Hospitals partially participating or not participating in OBI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This quality project will occur within the Obstetrics Initiative (OBI), a Blue Cross Blue Shield of Michigan (BCBSM)-funded collaborative of 68 Michigan hospitals dedicated to maternity care quality improvement. OBI's member hospitals constitute diverse maternity practice settings, ranging from urban to rural, academic to community, and high to low volume maternity units. OBI's quality initiative, "Bringing Our Patients COMFORT," will promote adoption of the COMFORT CPG across member hospitals. To the degree that OBI clinical champions share OBI initiative QI resources on their units, maternity clinicians staffing OBI hospitals will be exposed to these activities. To the degree that OBI hospitals adopt the COMFORT CPG, birthing populations at these sites will be exposed to guideline-concordant care.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Postpartum opioid prescribing - Rate | 18 months
  Rate of opioid prescribing within three days of discharge from the childbirth hospitalization
Postpartum opioid prescribing - Amount | 18 months
  Amount of opioid prescribed (oral morphine equivalent) within three days of discharge from the childbirth hospitalization

SECONDARY OUTCOMES:
Refill opioid prescribing | 18 months
  Rate of refill opioid prescriptions in the 30 days after discharge from the childbirth hospitalization
High-risk opioid prescribing | 18 months
  Prescription >50 oral morphine equivalents, overlapping opioid/benzodiazepine prescribing, and overlapping opioid prescriptions, all in the 30 days after discharge from the childbirth hospitalization

OTHER OUTCOMES:
Patient-reported outcomes | 21 months
  Pain intensity in the first week after childbirth, opioid consumption in the first week after discharge from the childbirth hospitalization, and satisfaction with pain management after discharge from the childbirth hospitalization
Implementation outcomes - reach | 21 months
  Characteristics of patients receiving guideline-concordant care vs. all patients
Implementation outcomes - adoption | 21 months
  Characteristics of responding hospitals and providers vs. all hospitals and providers
Implementation outcomes - feasibility | 21 months
  Provider perceptions of implementation intervention feasibility, as assessed by surveys and/or qualitative methods
Implementation outcomes - acceptability | 21 months
  Provider perceptions of implementation intervention acceptability, as assessed by surveys and/or qualitative methods
Implementation outcomes - appropriateness | 21 months
  Provider perceptions of implementation intervention appropriateness, as assessed by surveys and/or qualitative methods
Implementation outcomes - fidelity | 21 months
  Fidelity to assigned intervention, as measured via Coordinating Center administrative records (e.g., website downloads, training attendance, coaching call attendance)
Implementation outcomes - potential mechanisms of implementation | 21 months
  Qualitatively assessed indicators of potential mechanisms of effect, factors affecting implementation, and local adaptations to the guideline
Implementation outcomes - costs of delivering implementation | 21 months
  Coordinating Center costs for offering implementation support

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Moniz MH, Kilbourne AM, Peahl AF, Waljee JF, Cocroft S, Simpson C, Kane Low L, Bicket MC, Englesbe MJ, Stout MJ, Gunaseelan V, Bourdeau A, Hu M, Miller C, Smith SN. Can theory-driven implementation interventions help clinician champions promote opioid stewardship after childbirth? Protocol for a pragmatic implementation study. Front Glob Womens Health. 2025 Mar 14;6:1504511. doi: 10.3389/fgwh.2025.1504511. eCollection 2025. PMID 40160195